CLINICAL TRIAL: NCT05074069
Title: PelvEx 7: A Review of Functional and Surgical Outcomes of Gynaecological Reconstruction in the Context of Pelvic Exenteration
Brief Title: A Review of Functional and Surgical Outcomes of Gynaecological Reconstruction in the Context of Pelvic Exenteration
Status: Completed | Type: Observational
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Des Winter, Professor Desmond C Winter, St Vincent's University Hospital, Ireland
Other Study IDs: PelvEx 7
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Cancer
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neovaginal reconstruction: Neovaginal reconstruction post-vulvovaginal resection
  Interventions: Procedure: Gynaecological reconstruction
- Flap Reconstruction: Flap closure of perineal defect post-gynaecological organ resection
  Interventions: Procedure: Gynaecological reconstruction
- No reconstruction/Primary closure: Primary closure of defect post-multivisceral, gynaecological organ-involving, resection

INTERVENTIONS:
Procedure: Gynaecological reconstruction — Methods of vulvovaginal reconstruction, e.g. flap formation, neovagina formation
  Groups: Flap Reconstruction; Neovaginal reconstruction

SUMMARY:
Patients with locally advanced pelvic malignancy undergo radical procedures, necessitate organ reconstruction. Little is known about the preferred methods of gynaecological organ reconstruction in the context of pelvic exenteration. This review aims to identify which methods are commonly used and what outcomes are associated with each technique in order to further guide future practice.

DETAILED DESCRIPTION:
The mainstay of treatment for patients with locally advanced pelvic malignancy is radical surgical excision combined, with (neo)adjuvant chemoradiotherapy where appropriate. The primary objective is to obtain a negative resection margin (R0) in order to achieve long-term survival. Centralisation of care and refinements in surgical technique have enabled surgeons specializing in advanced pelvic oncology to embark upon more aggressive approaches to accomplishing an R0 resection.

With improved oncological outcomes has come an increased focus on quality-of-life (QoL), functional sequelae and patient experience and survivorship. Adequate experience and proficiency with reconstructive techniques has become one of the key components for surgeons practicing in pelvic oncology. Reconstructive procedures should be undertaken with the goals of improving wound healing, reducing morbidity and restoring anatomic form and function. These factors are of utmost importance in the context of pelvic exenteration, where wound complications are prevalent as a result of a larger pelvic dead space and the potential for contamination. Adverse impact on sexual function following pelvic surgery is also common where the autonomic nerves are involved. This is further compounded by the need to resect part or all of the vulvovaginar complex as part of an extirpative procedure, with resultant declines in QoL and overall psychosexual wellbeing.

A number of methods have been proposed for reconstruction of the pelvic floor and vulva/vagina in females, including skin grafting, skin flaps, fasciocutaneous and myocutaneous flaps, as well as the formation of a neovagina in specific circumstances. Thereis a paucity of data with regard to the optimal approach to gynaecological organ reconstruction, with the majority of the literature referring to single-centre, retrospective series. This review sought to assess the preferred methods for gynaecological reconstruction at an international level, the clinical and technical particulars leading to the choice of each method and the short-term outcomes associated with each technique.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or recurrent pelvic cancer (all subtypes - Rectal, Urological, Gynae, Sarcome)
* Aged over 18 years
* Undergoing a multi-visceral extended pelvic resection and requiring gynaecological reconstruction at the time of index operation
* Time period: 1st July 2016 - 31st July 2021

Exclusion Criteria:

* Strong evidence of metastatic or peritoneal disease
* No histological evidence of gynaecological organ involvement
* Procedure not carried out with curative intent
* Insufficient patient follow-up (Minimum of 30 days)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynaecological organ reconstruction only.
Study Population: Patients over 18 years of age who have undergone pelvic exenteration/multi-visceral resection with gynaecological organ reconstruction for a locally advanced pelvic malignancy in a participating PelvEx centre between July 2016 and July 2021.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | July 2016 - July 2021
  Number of patients experiencing short-term (up to 30 days postoperatively) morbidity
Gynaecological Reconstruction | July 2016 - July 2021
  Number of patients with each method of reconstruction
Perineal wound complications | July 2016 - July 2021
  Number of patients with superficial wound infections, abscess, dehiscence by type of reconstruction

SECONDARY OUTCOMES:
Dyspareunia | July 2016 - July 2021
  Dyspareunia
Return to intercourse | July 2016 - July 2021
  Return to intercourse
Pelvic pain | July 2016 - July 2021
  Chronic pelvic pain by type of reconstruction
Histological outcomes | July 2016 - July 2021
  Radicality of resection, e.g. R0, R1 or R2, and histological subtypes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Patients will be identified by a key from the nominated study coordinator from each site, with no individual or identifiable data to be shared between researchers.

REFERENCES:
- [Derived] PelvEx Collaborative. A review of functional and surgical outcomes of gynaecological reconstruction in the context of pelvic exenteration. Surg Oncol. 2024 Feb;52:101996. doi: 10.1016/j.suronc.2023.101996. Epub 2023 Nov 22. PMID 38096764